CLINICAL TRIAL: NCT04908969
Title: Internet-based Cognitive Behavioral Therapy for Chronic Tic Disorder and Tourette's Disorder: a Feasibility Trial
Acronym: TICNET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Christian Rück, Professor, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-00479
Record Dates: First submitted 2021-05-26; First posted 2021-06-01 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Chronic Tic Disorder; Tourette Syndrome
MeSH Terms: conditions — Tic Disorders; Tourette Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Internet-delivered Cognitive Behavior Therapy for Chronic Tic Dosorder/Tourette Disorder — The treatment will be provided through a secure internet platform designed for internet-administered treatments (BASS-4). In the treatment, the patient works through modules of self-help material, each ending in a short quiz with questions about the material. The treatment is supported by a therapist through text-based communication via the platform as well as occasional phone calls when needed. The central component in the treatment is exposure and response prevention (ERP). In ERP, the patient exposes her/himself to situations that trigger premonitory urges (a type of bodily sensation that precede the tic) while practicing to resist the tic. By doing this systematically and repeatedly, the patient gradually learns how to tolerate the premonitory urges and increase the ability to control and resist doing tics. Beyond ERP the treatment consists of other components such as applied relaxation, counter-movements and interventions to decrease stressors in the patient's everyday life.

SUMMARY:
Tic disorders, including Tourette's Disorder (TD) and Chronic Motor or Vocal Tic Disorder (CTD), are neurodevelopmental motor disorders characterised by motor and/or vocal tics. TD/CTD are impairing conditions with onset during childhood that often persist into adulthood. Behaviour therapy (BT) is an effective treatment for TD/CTD and is recommended as a first-line intervention in both in children and in adults. However, most adults with TD/CTD do not have access to BT due to a lack of trained professionals and geographical barriers. The objective of the study is to adapt and extend existing face-to-face BT treatment protocols for adults with TD/CTD to an internet-delivered format and evaluate its feasibility and preliminary efficacy. A total of 30 adult TD/CTD adult patients deemed eligible for the study through the recruitment process involving both psychologist and physician assessment will be enrolled in the project. The 8-modues treatment program, mainly based on exposure with response prevention with addition of other techniques will be made available for the participants in a secure treatment platform. The participants will keep in touch with a therapist using two-ways written communication in the same platform. The therapist's role will be to introduce the treatment and its modules, give feedback on the homework assignments and open the new modules as well as monitor the participants psychiatric symptoms and activity in the plattform. The measures will include tic severity secifically and disease severity in general, anxiety and depression symptoms, quality of life, treatment credibility and therapeutic alliance. The measures will be administrated at baseline, min- and post-tretment, as well at 3 and 12 months follow-up. Upon completion, this project will be the first crucial step towards the implementation of internet-delivered behaviour therapy (I-BT) for adults with TD/CTD in regular health care.

DETAILED DESCRIPTION:
Background

TS (Tourette Syndrome) is characterized by multiple motor tics and one or more vocal tics that have persisted for at least one year since initial onset, whereas in Chronic Motor or Vocal Tic Disorder (CTD) either motor or vocal tics are present, but not both, during at least one year (1). It is a childhood-onset disorder that affects more boys than girls (4:1 ratio) with a prevalence of about 1% in children (2), of which a substantial proportion continue to experience impairing tics into adulthood (3,4,5). TS/CTD are associated with reduced quality of life (6), lower educational attainment (7), and increased risk for cardiovascular and metabolic disorders (8). Notably, individuals with TD/CTD have a four-fold increased risk of death by suicide and the risk is highest for those whose tics persist into adulthood (9). Thus, effective interventions and appropriate follow-up are crucial to prevent undesirable health consequences and societal costs.

Evidence-based treatments for Tourette's Disorder and Chronic Tic Disorder

Historically, the most common treatment for TS/CTD has been pharmacotherapy, specifically antipsychotics. However, pharmacological treatments are modestly efficacious in reducing tics and often have undesirable side effects such as tiredness or long-term metabolic problems (10). Non-drug treatments for TS/CTD are therefore attractive alternatives. Behavioural treatments acknowledge that tics have a biological origin but that their expression is influenced by contextual variables: feelings, sensations, situations or other triggers that occur before tics. CBT focuses on modifying environmental factors that influence tic severity and teaches patients specific skills they can use to better manage their tics (11). CBT for tics generally includes two main elements. First, the patient learns how to detect their tics on a daily basis. Secondly, the patient learns how to resist the tics. CBT for TS/CTD has shown to be effective against waiting list (12) and against an active control group (13-16), with sustained results up to one year after treatment completion (17, 18). Expert guidelines in Europe and elsewhere recommend CBT as the first-line treatment for TS/CTD (17, 18).

Preferred treatments are not available

Surveys among young people with tics and their parents indicate that cognitive behavioural therapy is their preferred treatment option (19). However, this intervention is not widely available for TS/CTD (20). Thus, despite patient preferences and the problematic side effects of drugs, the vast majority of TS/CTD patients in Sweden receive only medication to treat their tics. Members of our team conducted an epidemiological study looking at all patients diagnosed with TS or CTD (n=6,979) in Sweden and found that over 75% of them received at least one drug, and over 70% were on at least two types of drugs. Moreover, prescription of anxiolytics, hypnotics/sedatives, ADHD drugs, and atypical antipsychotics increased over the 8-year study period (21).

In sum, expert therapists trained to treat TS/CTD with CBT in Sweden are lacking. Even in Stockholm County, it is our clinical experience that many adult patients with TS/CTD have trouble finding the appropriate expertise when seeking treatment in primary care, neurology, or psychiatry.

A remote cognitive behavioural intervention for adults with Tourette Syndrome

There has been an increase in uptake of information and communication technology within health care in recent years. One such innovation is to provide the treatment online instead of face-to-face. In internet-delivered psychological treatments, the treatment is provided in the form of self-help texts, homework assignments, and worksheets for the patient to fill in online. An identified therapist provides support and guidance throughout treatment via a built-in messaging system. Internet-delivered treatments is a burgeoning research field where Sweden is at the forefront of international development (22). Internet-delivered treatments have been developed and evaluated by our research team for many psychiatric conditions, including disorders related to TS/CTD, such as obsessive-compulsive disorder (OCD) and body dysmorphic disorder (BDD) (23-26). Internet-delivered treatments have consistently shown comparable effects to traditional face-to-face therapies (27) while requiring less therapist time per patient and being delivered remotely, thus being cost-effective for health care and accessible to patients (28). Preliminary results suggest that videoconferencing (29) and I-CBT (30) are feasible options for children with TS/CTD, but there are no such treatments available to adults with TS/CTD.

Research questions

There is an urgent need to disseminate evidence-based treatments for adults with TS and CTD. Internet-delivered cognitive behavioural therapy (ICBT) for TD/CTD will be a feasible, acceptable, and safe method to deliver evidence-based treatment for adults with TS/CTD. We also hypothesize that I-CBT will show preliminary efficacy in reducing tic severity in this population.

Methods

Study design

The aim of the project will be to carry out a pilot trial to evaluate the feasibility, acceptability, safety, and efficacy of the internet-delivered treatment for TS/CTD. We also aim to further refine the treatment based on feedback from participants and therapists involved in the trial. Furthermore, information obtained from this feasibility trial will allow us to investigate key design and methodological issues to inform the protocol of a subsequent full scale randomised controlled trial. Specifically, the generated within participant data will be critical to perform a power analysis for a more definitive trial (see power analysis section).

The study design and outcomes will be registered online at ClinicalTrials.gov prior to inclusion of the first participant. We will also upload the scripts used for statistical analyses to an online repository (such as the Open Science Framework or Github).

Outcome measures

Feasibility measures: Feasibility will be assessed according to the RE-AIM framework (reach, effectiveness, adoption, implementation, maintenance) (33). Reach will be measured by looking at the percentage eligible/excluded, reasons for refusal or exclusion.

Efficacy measures: Unless specified otherwise, all outcome measures will be administered at baseline, post-treatment (primary end-point), 3-month follow-up, 6-month follow-up, and 12-month follow-up. Primary outcome measure: YGTSS TTSS. Secondary disorder-specific outcomes: YGTSS Impairment scale, Adult Tic Questionnaire (weekly). Functioning and quality of life measures: The Clinical Global Impression - Severity (CGI-S) and Clinical Global Impression - Improvement (CGI-I) Scales will be used to assess overall clinical severity and consequent treatment response (scores of "very much improved" (1) or "much improved" (2) will define treatment response according to previous trials in tic disorders (14, 16). In addition, Global Assessment of Functioning (GAF), Sheehan Disability Scale (SDS), EuroQol 5-dimensions (EQ-5D), Gilles de la Tourette Syndrome Quality of Life Scale (QTS-QoL) will be used to evaluate functioning and quality of life. Depressive symptoms: MADRS-S will be administered weekly to follow depressive symptoms during treatment.

Procedure

Patients with TS/CTD will be recruited through our clinic (OCD-programmet) as well as through self-referral. Information about the study will be communicated to patient associations (such as OCD-förbundet and Attention), health centers, psychiatric outpatient clinics, internal referral systems (remissportal) as well as advertised in the media and in social media. Self-referral will be made available through an internet website constructed for the study. The website will contain information about the study, the research group, and contact information. Screening: Self-referred participants will go through a telephone screening containing information about the study and an assessment of inclusion and exclusion criteria. If the presumptive participant is deemed fit for inclusion, they will be scheduled for a visit with a study clinician. Patients that are recruited through internal referral systems will not go through the screening procedure but will be scheduled for a visit with a study clinician. Assessment: Potential participants will be assessed face to face at our clinic in Stockholm for eligibility to participate (see inclusion and exclusion criteria above) by a study clinician. The assessment includes an assessment if the participant fulfil the diagnostic criteria of a TS/CTD diagnosis based on a review of medical history and the DSM-5 diagnostic criteria. The YGTSS will be administered to establish symptom severity. A semi-structured clinical psychiatric interview (the Mini-International Neuropsychiatric Interview; MINI), as well as the SCID-1 section for OCD and related disorders (OCD, BDD, tricho- and dermatillomania, hoarding disorder) will be administered in order to assess psychiatric comorbidities. This routine corresponds to the regular diagnostic assessment at the clinic. Patients suitable for study participation will be given information about the study and asked to sign a form giving their informed consent to participate in the study. Participants will initiate treatment within a week and begin by filling in self-report measures on the internet (listed under Efficacy measures, above). Patients who decline participation in the study will be offered regular treatment at the clinic or, depending on the individual's needs, be referred to other clinical services.

Treatment

Interventions: As described above, the treatment protocol will be adapted from existing validated protocols for face-to-face treatment and remote delivery (12-16, 30).

The treatment will be provided through a secure internet platform designed for internet-administered treatments (BASS-4). The platform has been studied extensively and is currently a part of the Swedish public health care services. In the treatment, the patient works through modules of self-help material, each ending in a short quiz with questions about the material. The treatment is supported by a therapist through text-based communication via the platform as well as occasional phone calls when needed. The central component in the treatment is exposure and response prevention (ERP). In ERP, the patient exposes her/himself to situations that trigger premonitory urges (a type of bodily sensation that precede the tic) while practicing to resist the tic. By doing this systematically and repeatedly, the patient gradually learns how to tolerate the premonitory urges and increase the ability to control and resist doing tics. Beyond ERP the treatment consists of other components such as applied relaxation, counter-movements and interventions to decrease stressors in the patient's everyday life.

Therapist training, supervision, and quality control

Therapists will be licensed clinical psychologists, psychologists in training or fifth-year clinical psychology students under supervision. As all communication with the patients is stored in the platform, continuous monitoring and supervision is possible and will be provided by the study coordinator to ensure adherence. All assessors will be trained on the use of the primary outcome measure, the YGTSS (32) using case examples, and inter-rater reliability scores will be obtained. The study is approves by the Ethical Review Authority. The trial will be conducted in accordance with Good Clinical Practice (GCP) and results will be reported in accordance with the CONSORT statement for non-pharmacological trials.

Statistical analysis

Power calculation

Given a standardized (Cohen's d) within-group effect size of 0.5 to 1 in previous research of remote therapy for TS/CTD (30), we aim to recruit 30 participants in order to be able to detect an effect size of d = 0.7, allowing for a 20% dropout (90% power, alpha 0.05). The primary outcome analysis will also inform the power analyses of a future large-scale randomised controlled trial via the variance of intercept, fixed effects, random effects, and residual variance for the YGTSS in the mixed effects model. These estimates will help us select the appropriate number of participants to make the results from the randomised controlled trial informative and useful.

Outcome analyses

The primary and secondary outcome measures will be evaluated using mixed-effects linear regression models with a fixed effect of time, as well as random intercept and random slope specifications for each individual. Within-group effect sizes will be calculated using Cohen's d by dividing the mean change between the time-points by the pooled standard deviation of that measure at pre-treatment. To maximize replicability and transparency, all statistical code will be published in public repositories.

ELIGIBILITY:
Inclusion Criteria:

The participant should

1. be 18 years of age or older,
2. fulfill diagnostic criteria for Tourette's Disorder (from now on referred to as Tourette Syndrome; TS) or Persistent (Chronic) Motor or Vocal Tic Disorder (CTD) according to the DSM-5 diagnostic criteria,
3. have Total Tic Severity Score [TTSS] of >15, or >10 for individuals with motor or vocal tics only, in the past week as measured by the Yale Global Tic Severity Scale (YGTSS) (31) ,
4. be able to read and communicate in Swedish and
5. have regular access to a computer connected to the internet, sufficient technical skills to use the treatment platform, as well as a mobile phone to receive SMS.

Exclusion Criteria:

1. organic brain disorders, intellectual disability, psychosis, bipolar disorder, autism spectrum disorder, anorexia nervosa, or substance use disorders,
2. acute psychiatric problems such as severe depression or suicidal risk needing immediate psychiatric care,
3. severe tics causing immediate risk to the patients or others and requiring urgent medical attention,
4. previous CBT for tics of a minimum of 8 sessions with a qualified therapist within 12 months prior to assessment,
5. simultaneous psychological treatment for TS or CTD
6. initiation or adjustment of medication for tics within the last two months prior to assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2023-06-23 (Estimated); Study Completion 2023-08-23 (Estimated)

PRIMARY OUTCOMES:
Yale Global Tic Severity Scale (YGTSS) | For the primary outcome: change between baseline and three months follow-up with one additional in-between measures at post-tretment. Two additional follow-up measures at 6- and 12-months.
  The YGTSS is made up of a semi-structured interview, followed by a questionnaire where individuals are asked to rate the severity of their Tic symptoms (both motor and vocal) in domains such as: number, frequency, intensity, complexity, and interference. There is also an impairment scale, where the individual rates how the Tic impacts on their daily life and activities. The Total Tic Severity Score has a range of 0-50, and the Global Severity Score has a range of 0- 100. A higher score on all scales suggests a more severe Tic, or a greater impact the Tic has on the person's life. Only the total tic severity core will be used as the primary outcome.

SECONDARY OUTCOMES:
Yale Global Tic Severity Scale (YGTSS) - impairment scale | Change between baseline and three months follow-up with one additional in-between measure at post-tretment. Two additional follow-up measures at 6- and 12-months.
  The YGTSS is made up of a semi-structured interview, followed by a questionnaire where individuals are asked to rate the severity of their Tic symptoms (both motor and vocal) in domains such as: number, frequency, intensity, complexity, and interference. There is also an impairment scale, where the individual rates how the Tic impacts on their daily life and activities. The Total Tic Severity Score has a range of 0-50, and the Global Severity Score has a range of 0- 100. A higher score on all scales suggests a more severe Tic, or a greater impact the Tic has on the person's life. The impairment scale will be used as a secondary outcome measure.
Clinical Global Impression (CGI) | Change between baseline and three months follow-up with one additional in-between measure at post-tretment. Two additional follow-up measures at 6- and 12-months.
  The Clinical Global Impression - Severity (CGI-S) and Clinical Global Impression - Improvement (CGI-I) Scales will be used to assess overall clinical severity and consequent treatment response (scores of "very much improved" (1) or "much improved" (2) will define treatment response according to previous trials in tic disorders.
Global Assessment of Functioning (GAF) | Change between baseline and three months follow-up with one additional in-between measure at post-tretment. Two additional follow-up measures at 6- and 12-months.
  GAF-scale measures how much a person's symptoms affect their everyday life on a scale of 0 to 100, with higher score indicating better functioning.
Sheehan Disability Scale (SDS) | Change between baseline and three months follow-up with one additional in-between measure at post-tretment. Two additional follow-up measures at 6- and 12-months.
  SDS assesses functional impairment in three domains: work/school, social and family life. Each domain is scored on a scale from 0 to 10 with higher scores indicating more severe impairment. The total score ranges from 0 t 30.
EuroQol 5-dimensions (EQ-5D) | Change between baseline and three months follow-up with one additional in-between measure at post-tretment. Two additional follow-up measures at 6- and 12-months.
  EQ-5D evaluates the generic quality of life. In covers 5 dimensions: mobility, self-care, usual activity, pain/discomfort, anxiety/depression that are rated on a 5-point likert scale from not having any impairment to having a severe impairment.
Gilles de la Tourette Syndrome Quality of Life Scale (QTS-QoL) | Change between baseline and three months follow-up with one additional in-between measure at post-tretment. Two additional follow-up measures at 6- and 12-months.
  QTS-QoL is a syndrom-specific quality of life scale with 27 items scored on a 5-point likert scale from no problems to very severe problems.The total score ranges from 0 to 108 with higher score indicating more severe problems.
Montgomery-Asberg Depression Rating Scale (MADRS) | Weekly measurements starting a baseline through post-tretment. Two additional follow-up measures at 6- and 12-months.
  MADRS is a 9-item depressive symptoms scale where the symptoms are assessed on a 7-point likert scale from no symtoms to very high severity. The total score ranges from 0 to 54 with higher score indicating more severe problems.

OTHER OUTCOMES:
Internet Intervention Patient Adherence Scale for Guided Internet-Delivered Behavioural Interventions (iiPAS) | Administered at mid- and post-treatment.
  The iiPAS is a 5-item, clinician-rated measure of patient adherence to internet-delivered behavioral interventions. The 5 items are rated by treating clinicians and cover 5 central aspects of adherence: the patient's work pace, engagement, communication with the clinician, motivation for change, and login frequency. The clinicians assess each domain on a 5-point likert scale (scored 0-4), with a total score ranging between 0-20 where higher score indicates higher treatment adherence.
Credibility/Expectancy Questionnaire (CEQ) | In the 4th week of the treatment.
  The CEQ is a 5-item measure of the treatment's credibility and the patients' expectations. The patients assess each domain on a 11-point likert scale (scored 0-10), with a total score ranging between 0-50 where higher score indicates higher credibility and higher expectations.
Working Alliance Inventory Short-Revised (WAI-SR) | In the 4th week of the treatment.
  The WAI-SR is a 12-item measure of the patient's experience of their working alliance with the therapist. The patients assess each item on a 7-point likert scale (scored 0-6), with a total score ranging between 0-72 where higher score indicates higher better working alliance according to the patient.
Client Satisfaction Questionnaire (CSQ-8) | At post-treatment.
  The CSQ is an 8-item measure of the patient's satisfaction with the treatment. The patients assess each domain on a 4-point likert scale (scored 0-3), with a total score ranging between 0-24 where higher score indicates higher satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- OCD-clinic, Psykiatri Sydväst, Huddinge hospital, Huddinge, Sweden